CLINICAL TRIAL: NCT01844778
Title: An Open-label, Crossover, Interventional Phase IV Study to Compare the Ease of Use of TIP With Nebulized TIS and Nebulized COLI for the Treatment of Pulmonary Pseudomonas Aeruginosa (P.a) in Patients With Cystic Fibrosis
Brief Title: Ease of Use and Microbial Contamination of Tobramycin Inhalation Powder (TIP) Versus Nebulised Tobramycin Inhalation Solution (TIS) and Nebulised Colistimethate (COLI)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CTBM100C2403; 2012-001565-33 (EudraCT Number)
Record Dates: First submitted 2013-04-29; First posted 2013-05-01 (Estimated); Results first posted 2016-05-24 (Estimated); Last update posted 2016-07-27 (Estimated); Status verified 2016-07

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis, Pseudomonas aeruginosa, FEV1, tobramycin inhalation powder, TOBI,; colistimethate; Cystic Fibrosis, Pseudomonas aeruginosa, FEV1, tobramycin inhalation powder, TOBI, colistimethate
MeSH Terms: conditions — Cystic Fibrosis; Pseudomonas Infections | interventions — colistinmethanesulfonic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- TIS/TIP (Active Comparator): During the first cycle of treatment, participants received nebulized TIS, 300 mg twice per day for 28 days followed by 28 days off-treatment. During the second cycle, participants received 112 mg (four 28 mg capsules) twice per day for 28 days followed by 28 days off-treatment.
  Interventions: Drug: Tobramycin Inhalation Powder; Drug: Tobramycin inhalation solution
- COLI/TIP (Active Comparator): During the first cycle, participants received nebulized COLI, 1 million or 2 million units twice or thrice per day (or the participant's usual dose and regimen) for 56 days (no off-treatment period) or 28 days on-treatment followed by 28 days off-treatment (cycling regimen), depending on local treatment guidelines. During the second cycle, participants received TIP, 112 mg (four 28 mg capsules) twice per day for 28 days followed by 28 days off-treatment.
  Interventions: Drug: Tobramycin Inhalation Powder; Drug: Colistimethate
- TIP/TIP (Active Comparator): During the first and second cycles, participants received TIP, 112 mg (four 28 mg capsules) twice per day for 28 days followed by 28 days off-treatment.
  Interventions: Drug: Tobramycin Inhalation Powder

INTERVENTIONS:
Drug: Tobramycin Inhalation Powder — Tobramycin Inhalation Powder was administered via TOBI® Podhaler (T-326 inhaler).
  Other Names: TIP
Drug: Tobramycin inhalation solution — Tobramycin inhalation solution was administered via nebuliser
  Other Names: TIS
  Arms: TIS/TIP
Drug: Colistimethate — Colistimethate was administered via nebuliser.
  Other Names: COLI
  Arms: COLI/TIP

SUMMARY:
The purpose of this interventional Phase IV study was to explore the ease of use of TIP and prevalence of microbial contamination of the T-326 Inhaler compared with TIS and colistimethate administered via nebuliser for the treatment of Cystic Fibrosis (CF) patients chronically infected with P. aeruginosa.

It was anticipated that the data from this study would provide clinicians with further guidance on the relative differences between the speed and ease of use of these treatments as well as useful information on the prevalence of microbial contamination of the inhalation devices in "real world" use.

DETAILED DESCRIPTION:
Patients who were on colistimethate (COLI), Tobramycin Inhalation Powder (TIP) or Tobramycin Inhalation Solution (TIS) were recruited for the study. They went through one treatment cycle on their usual inhaled antibiotic treatment, and were all transferred to TIP for the second treatment cycle. The primary endpoint was the total administration time of TIP vs TIS vs colistimethate, defined as the total time taken to prepare the delivery device and drug, administer the drug, and clean and disinfect the delivery device.

ELIGIBILITY:
Key Inclusion Criteria:

* Provide written informed consent, HIPAA authorization, and assent (as appropriate for minors) prior to the performance of any study-related procedure
* Confirmed diagnosis of Cystic Fibrosis (CF)
* Male and female patients 6 years of age or older at screening
* Forced Expiratory Volume in 1 second (FEV1) at screening (Visit 1) must be at least 25% and less than or equal to 90% of normal predicted values for age, sex, and height based on the NHANES III values (Hankinson, 1999) for patients 18 years of age or greater, and based on values from Wang (Wang 1993) for patients less than 18 years of age.
* Documented use of any of the nebulized antibiotics based on local practice:
* Tobramycin Inhalation Solution, colistimethate, or Tobramycin Inhalation Powder for at least 1 cycle within the last 6 months or
* Colistimethate continuous use for at least 8 weeks within the last 6 months This cycle of treatment (or continuous colistimethate treatment period) is in addition to the treatment cycle during which the subject is being screened.
* P. aeruginosa must be present in a sputum or deep cough throat swab culture or bronchoalveolar lavage (BAL) (only for BAL a threshold level of 10^3 CFU/mL is required) within 6 months prior to screening, and in the sputum or deep cough throat swab culture at screening or rescreening (Visit 1);

Key Exclusion Criteria:

* History of sputum culture or deep cough throat swab (or BAL) culture yielding Burkholderia cenocepacia complex within 2 years prior to prescreening or sputum culture yielding B. cenocepacia complex at screening (Visit 1)
* History of hearing loss or chronic tinnitus deemed clinically significant by the investigator
* Serum creatinine 176.8 μmol/L (2 mg/dL) or greater, blood urea nitrogen (BUN) 14.28 mmol/L (40 mg/dL) or greater, or an abnormal urinalysis defined as 2+ or greater proteinuria at screening
* Known local or systemic hypersensitivity to aminoglycosides
* Regularly receiving more than 1 class of inhaled antipseudomonal antibiotic
* Use of any investigational drug within 30 days or 5 half-lives, whichever is longer, prior to screening
* Signs and symptoms of acute pulmonary disease, e.g., pneumonia, pneumothorax
* Body mass index less than 12 kg/m2
* History of malignancy of any organ system, treated or untreated
* Clinically significant laboratory abnormalities (not associated with the study indication) at screening (Visit 1)
* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive human chorionic gonadotropin (hCG) laboratory test
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using effective methods of contraception during study treatment.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-08; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (21):
- Germany (4):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Tübingen
- Novartis Investigative Site, Galway, Ireland
- Spain (5):
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, Palma de Mallorca, Balearic Islands
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Madrid, Madrid
  - Novartis Investigative Site, Valencia, Valencia
- Switzerland (3):
  - Novartis Investigative Site, Basel, Switzerland
  - Novartis Investigative Site, Zurich, Switzerland
  - Novartis Investigative Site, Sankt Gallen
- United Kingdom (8):
  - Novartis Investigative Site, Southampton, Hampshire
  - Novartis Investigative Site, Penarth, Vale of Glamorgan
  - Novartis Investigative Site, Birmingham, West Midlands
  - Novartis Investigative Site, Bristol
  - Novartis Investigative Site, East Yorkshire
  - Novartis Investigative Site, Exeter
  - Novartis Investigative Site, Liverpool
  - Novartis Investigative Site, Newcastle upon Tyne

REFERENCES:
- [Derived] Greenwood J, Schwarz C, Sommerwerck U, Nash EF, Tamm M, Cao W, Mastoridis P, Debonnett L, Hamed K. Ease of use of tobramycin inhalation powder compared with nebulized tobramycin and colistimethate sodium: a crossover study in cystic fibrosis patients with pulmonary Pseudomonas aeruginosa infection. Ther Adv Respir Dis. 2017 Jul;11(7):249-260. doi: 10.1177/1753465817710596. PMID 28614995

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Each participant was assigned to 1 of 3 treatment arms, TIS/TIP, COLI/TIP, or TIP/TIP with the first treatment cycle based on the participant's usual antibiotic treatment. Then all participants were crossed-over to receive TIP for the second cycle of treatment.
Groups:
- TIS/TIP: During the first cycle of treatment, participants received nebulized TIS, 300 mg twice per day for 28 days followed by 28 days off-treatment. During the second cycle, participants received TIP 112 mg (four 28 mg capsules) twice per day for 28 days followed by 28 days off-treatment.
- COLI/TIP: During the first cycle, participants received nebulized COLI, 1 million or 2 million units twice or thrice per day (or the participant's usual dose and regimen) for 56 days (no off-treatment period) or 28 days on-treatment followed by 28 days off-treatment (cycling regimen), depending on local treatment guidelines. During the second cycle, participants received TIP 112 mg (four 28 mg capsules) twice per day for 28 days followed by 28 days off-treatment.
- TIP/TIP: During the first and second cycles, participants received TIP 112 mg (four 28 mg capsules) twice per day for 28 days followed by 28 days off-treatment.
Period: Overall Study
Arm/Group | TIS/TIP | COLI/TIP | TIP/TIP
Started | 14 | 28 | 18
Safety Set 1 (at Least 1 Dose, Cycle 1) | 14 | 28 | 18
Safety Set 2 (at Least 1 Dose, Cycle 2) | 12 | 25 | 15
Completed | 12 | 25 | 14
Not Completed | 2 | 3 | 4
Not completed — Protocol deviation | 0 | 1 | 2
Not completed — Withdrawal by Subject | 2 | 0 | 0
Not completed — Adverse Event | 0 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TIS/TIP | COLI/TIP | TIP/TIP | Total
Number analyzed (Participants) | 14 | 28 | 18 | 60
Age, Continuous [Mean (Standard Deviation); unit: Years] | 27.4 (6.82) | 28.4 (9.86) | 26.6 (7.25) | 27.6 (8.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 10 | 7 | 21
  Male | 10 | 18 | 11 | 39

OUTCOME MEASURES:

1. Primary Outcome: Mean Total Administration Time
Description: The mean total time for administration of TIP via T-326 inhaler versus the total time for administration of COLI or TIS was assessed from information entered by participants into an ediary during the last 7 days prior to the last dose of a cycle. The total time included the setup, preparation, administration and cleaning/disinfection time.
Time Frame: days 22 through 28 (cycle 1), days 78 through 84 (cycle 2)
Population: The full analysis set (FAS) was considered for this analysis. The FAS included participants who received at least 1 dose of treatment. Only participants (n), with non-missing mean total administration time of initial and second cycles, were analyzed.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | TIS/TIP | COLI/TIP | TIP/TIP
Number analyzed (Participants) | 14 | 28 | 18
minutes
  Cycle 1 (n=8,17,14) | 37.0 (22.06) | 16.4 (9.54) | 4.2 (2.02)
  Cycle 2 (n=10,16,11) | 5.0 (2.04) | 3.8 (1.70) | 3.4 (2.06)

2. Secondary Outcome: Change in P. Aeruginosa Sputum Density
Description: Sputum samples were sent to a central laboratory at the start and end of 2 treatment periods. The absolute change in the number of colony forming units (CFU) of Pseudomonas aeruginosa in sputum = the value of end of on/off treatment period of the cycle minus the pre-dose value at the start of that cycle. A negative change from baseline indicates improvement.
Time Frame: days 1, 28 (cycle 1); 57, 84, 112 (cycle 2)
Population: The FAS was considered and included participants who received at least 1 dose of treatment. Only participants (n), with values at the start and end of an on-treatment period ("on-treatment" change), and/or with values at the start of an on-treatment period and end of an off-treatment period ("off-treatment" change), were analyzed.
Measure: Mean (Standard Deviation); unit: log10 CFU/mL
Arm/Group | TIS/TIP | COLI/TIP | TIP/TIP
Number analyzed (Participants) | 14 | 28 | 18
log10 CFU/mL
  Cycle 1, on-treatment change (n=11,22,9) | -1.4 (1.85) | -0.6 (1.88) | -1.7 (2.87)
  Cycle 1, off-treatment change (n=10,20,8) | 0.2 (1.98) | -0.6 (2.36) | -0.2 (1.56)
  Cycle 2, on-treatment (n=9,16,5) | -0.9 (1.66) | -0.5 (1.65) | -1.6 (1.53)
  Cycle 2, off-treatment (n=9,18,5) | 0.0 (0.95) | 0.5 (2.55) | 0.0 (0.91)

3. Secondary Outcome: Number of Participants With Any Contaminated Delivery Device
Description: Devices used to administer the drugs (the T-326 inhaler and nebulisers) were swabbed for contamination testing at the start and end of each treatment cycle (or discontinuation visit if the participant withdrew). No assessments were required from the T-326 inhaler when participants started the treatment period (days 1 and 57). Microbial contamination was measured according to device type and the frequency of organism growth (light/ moderate/ heavy). All nebulisers (neb) used by the participants were analyzed, including those for inhaling other medications, like mucolytics.
Time Frame: days (d) 1, 28, 57, 84
Population: The FAS was considered for the analysis and included participants who had at least one dose of study treatment. Only participants (n), with an available culture from the delivery device, were analyzed.
Measure: Number; unit: Participants
Arm/Group | TIS/TIP | COLI/TIP | TIP/TIP
Number analyzed (Participants) | 14 | 28 | 18
Participants
  P. a biotype 2 - dry,d1,neb, moderate,(n=0,0,1) | NA — no contamination | NA — no contamination | 1
  A. baumannii,d1,neb,heavy,n=0,7,0 | NA — no contamination | 1 | NA — no contamination
  A. junii,d1,neb,moderate,n=0,7,0 | NA — no contamination | 1 | NA — no contamination
  A.lwoffi,d1,neb,light,n=0,7,0 | NA — no contamination | 2 | NA — no contamination
  H. parainfluenza,d1,neb,light,n=0,7,0 | NA — no contamination | 1 | NA — no contamination
  O. anthropic,d1,neb,heavy,n=0,7,0 | NA — no contamination | 1 | NA — no contamination
  P. fluorescens,d1,neb,light,n=0,7,0 | NA — no contamination | 1 | NA — no contamination
  P. putida,d1,neb,light,n=0,7,0 | NA — no contamination | 1 | NA — no contamination
  P. stutzeri,d1,neb,moderate,n=0,7,0 | NA — no contamination | 1 | NA — no contamination
  S.liquefaciens,d1,neb,light,n=0,7,0 | NA — no contamination | 1 | NA — no contamination
  S. multivorum,d1,neb,light,n=0,7,0 | NA — no contamination | 1 | NA — no contamination
  S. maltophilia,d1,neb,light,n=0,7,0 | NA — no contamination | 1 | NA — no contamination
  Acinetobacter species,d28,neb,light,n=0,6,0 | NA — no contamination | 1 | NA — no contamination
  C. indologenes,d28,neb,moderate,n=0,6,0 | NA — no contamination | 1 | NA — no contamination
  D. acidovorans,d 28,neb,light,n=0,6,0 | NA — no contamination | 1 | NA — no contamination
  P. fluorescens,d28,neb,light,n=0,6,0 | NA — no contamination | 2 | NA — no contamination
  S. paucimobilis,d28,neb,heavy,n=0,6,0 | NA — no contamination | 1 | NA — no contamination
  S. aureus,d28,neb,light,n=0,6,0 | NA — no contamination | 1 | NA — no contamination
  P. a biotype 2 - dry,d57,neb,light,n=1,0,0 | 1 | NA — no contamination | NA — no contamination
  S. aureus,d84,T-326,light,n=1,0,0 | 1 | NA — no contamination | NA — no contamination

4. Secondary Outcome: Minimum Inhibitory Concentration (MIC) - MIC50 and MIC90 Tobramycin Values
Description: MIC50/90 is the lowest concentration required to inhibit 50%/90% of the isolates tested. The MIC50/90 of a range of antibiotics for P.aeruginosa was determined at the start and end of each treatment cycle, and at the end of the off-treatment period of the second cycle.
Time Frame: days 1, 28, 57, 84, 112
Population: The FAS was considered for the analysis and included participants who had at least one dose of study treatment. Only participants (n), with values on a given day, were analyzed for that day. The number of isolates tested = m.
Measure: Number; unit: ug/mL
Arm/Group | TIS/TIP | COLI/TIP | TIP/TIP
Number analyzed (Participants) | 14 | 28 | 18
ug/mL
  MIC50: Day 1, n=14,27,18; m=27,51,29 | 2 | 2 | 2
  MIC50: Day 28, n=13,23,13; m=25,46,21 | 2 | 2 | 2
  MIC50: Day 57, n=11,19,15; m=23,34,24 | 4 | 4 | 2
  MIC50: Day 84, n=12,17,11; m=25,29,18 | 4 | 4 | 2
  MIC50: Day 112, n=12,19,12; m=24,33,19 | 2 | 2 | 1
  MIC90: Day 1, n=14,27,18; m=27,51,29 | 256 | 16 | 64
  MIC90: Day 28, n=13,23,13; m=25,46,21 | 256 | 16 | 64
  MIC90: Day 57, n=11,19,15; m=23,34,24 | 64 | 16 | 64
  MIC90: Day 84, n=12,17,11; m=25,29,18 | 512 | 32 | 64
  MIC90: Day 112, n=12,19,12; m=24,33,19 | 32 | 32 | 32

5. Secondary Outcome: Number of Participants With Post-inhalation Bronchospasm
Description: Bronchospasm was defined as the relative decrease of 20% or more in forced expiratory volume in 1 second (FEV1) percent predicted from pre-dose to 15 to 45 minutes post-dose.
Time Frame: days 1, 28, 57, 84
Population: The FAS was considered for the analysis and included participants who had at least one dose of study treatment. Only participants (n), with values on a given day, were analyzed for that day.
Measure: Number; unit: Participants
Arm/Group | TIS/TIP | COLI/TIP | TIP/TIP
Number analyzed (Participants) | 14 | 28 | 18
Participants
  Day 1, n=8,17,14 | 0 | 1 | 0
  Day 28, n=6,19,14 | 0 | 1 | 0
  Day 57, n=10,22,13 | 0 | 0 | 1
  Day 84, n=8,14,10 | 0 | 0 | 0

ADVERSE EVENTS:
Groups:
- TIS/TIP - Cycle 1: During the first cycle of treatment, participants received nebulized TIS, 300 mg twice per day for 28 days followed by 28 days off-treatment.
- TIS/TIP - Cycle 2; COLI/TIP - Cycle 2: During the second cycle, participants received TIP 112 mg (four 28 mg capsules) twice per day for 28 days followed by 28 days off-treatment.
- COLI/TIP - Cycle 1: During the first cycle, participants received nebulized COLI, 1 million or 2 million units twice or thrice per day (or the participant's usual dose and regimen) for 56 days (no off-treatment period) or 28 days on-treatment followed by 28 days off-treatment (cycling regimen), depending on local treatment guidelines.
- TIP/TIP - Cycle 1; TIP/TIP - Cycle 2: During the first and second cycles, participants received TIP 112 mg (four 28 mg capsules) twice per day for 28 days followed by 28 days off-treatment.
- Overall TIP Cycle 2: During the second cycle, each treatment group received TIP 112 mg (four 28 mg capsules) twice per day for 28 days followed by 28 days off-treatment.
Arm/Group | TIS/TIP - Cycle 1 | TIS/TIP - Cycle 2 | COLI/TIP - Cycle 1 | COLI/TIP - Cycle 2 | TIP/TIP - Cycle 1 | TIP/TIP - Cycle 2 | Overall TIP Cycle 2
Serious Adverse Events (participants affected / at risk) | 3/14 | 3/12 | 9/28 | 3/25 | 3/18 | 2/15 | 8/52
Other Adverse Events (participants affected / at risk) | 5/14 | 6/12 | 13/28 | 12/25 | 10/18 | 10/15 | 28/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TIS/TIP - Cycle 1 (N=14) | TIS/TIP - Cycle 2 (N=12) | COLI/TIP - Cycle 1 (N=28) | COLI/TIP - Cycle 2 (N=25) | TIP/TIP - Cycle 1 (N=18) | TIP/TIP - Cycle 2 (N=15) | Overall TIP Cycle 2 (N=52)
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Faecaloma (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bile duct stenosis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Biliary tract disorder (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fungal infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 3 | 3 | 6 | 3 | 2 | 0 | 6
Influenza (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Acoustic stimulation tests abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Forced expiratory volume decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Pulmonary function test decreased (Investigations) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TIS/TIP - Cycle 1 (N=14) | TIS/TIP - Cycle 2 (N=12) | COLI/TIP - Cycle 1 (N=28) | COLI/TIP - Cycle 2 (N=25) | TIP/TIP - Cycle 1 (N=18) | TIP/TIP - Cycle 2 (N=15) | Overall TIP Cycle 2 (N=52)
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Distal intestinal obstruction syndrome (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Odynophagia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Influenza like illness (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Malaise (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 2
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1
Bile duct stone (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 2 | 1 | 5 | 6 | 0 | 1 | 8
Influenza (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 3 | 0 | 2 | 3 | 3
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Tongue fungal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 1
Tracheobronchitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vulvovaginal candidiasis (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 1
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Forced expiratory volume decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Glucose urine present (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Liver function test abnormal (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 1
Aphonia (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1
Burning sensation (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 3 | 3 | 3
Lethargy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 2 | 0 | 2 | 2 | 3
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 2 | 2 | 0 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Prolonged expiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 3 | 2 | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 2
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.